CLINICAL TRIAL: NCT07003659
Title: The Effects of a Tele-Yoga Program on University Students With Musculoskeletal Pain and Low Levels of Physical Activity
Brief Title: Tele-Yoga for Inactive Students With Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZY-2025
Record Dates: First submitted 2025-05-15; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Telerehabilitation; Yoga; University Students; Anxiety; Stress
Keywords: yoga; telerehabilitation; university students; anxiety; stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Group (Active Comparator): The yoga program was applied to the exercise group via video conference method as a group-based supervised standardized tele-rehabilitation program that allows individuals to perform their exercises in their own environment 3 days a week for 4 weeks. The tele-yoga program was applied as a Hatha yoga session of approximately 30 minutes consisting of yogic breathing exercises pranayama, asana practices expressing yoga poses and 10 minutes of meditation practice.
  Interventions: Other: Tele-Yoga
- Control Group (No Intervention): The control group did not receive any exercise program or therapeutic intervention

INTERVENTIONS:
Other: Tele-Yoga — This program consisted of diaphragmatic breathing, pranayama techniques consisting of nadi sodhana and ujjai, yoga poses consisting of sukhasana, bharadvajasana, marjaryasana - bitilasana, bhujaganasana, salabhasana, kapotasana, hasta uttanasana, virabhadrasana, adho mukha svanasana, bhujangasana. The exercises were carried out in a way that they would be followed up with an exercise diary in which they would take notes on continuing these exercises throughout the tele-yoga practice period, and reminder messages for the exercises were sent by the researchers to the WhatsApp group opened with the participants who participated in the study and were included in the exercise group.
  Other Names: yoga
  Arms: Tele-Yoga Group

SUMMARY:
Objective:

This study aimed to investigate the effects of a tele-yoga program on pain, functionality, anxiety, stress, and sleep quality in university students with musculoskeletal pain and low levels of physical activity.

Methods:

A total of 56 university students participated in the study (tele-yoga group: n=31; control group: n=25). The tele-yoga group received a standardized, supervised group-based tele-rehabilitation program delivered via videoconferencing, three times per week for four weeks. Participants performed the exercises in their own environments. No exercise intervention was applied to the control group. The same assessment protocol was conducted before and after the intervention in both groups.

DETAILED DESCRIPTION:
Musculoskeletal pain is a common pain in society and individuals experience pain in certain areas at certain times of their lives. Musculoskeletal pain is related to learned posture and habits, and it can be said that musculoskeletal pain occurring at older ages is also related to pain experienced at an early age. Musculoskeletal pain occurring in young adults may develop due to any organic pathology of neoplastic, inflammatory, infectious origin, and in the vast majority of cases, it develops due to factors such as posture and working conditions. In various studies conducted on the subject, it has been determined that gender, the grade studied, the department's computer use, the load carried by students, the daily sitting time, academic stress and exercise habits are effective in the formation of musculoskeletal pain experienced at an early age.Pain, the earliest symptom of musculoskeletal problems, is defined as an unpleasant sensory and emotional experience associated with existing or potential tissue damage. Emotional, behavioral and cognitive effects increase in long-term pain. It is stated that anxiety, one of these effects, is associated with many physical and psychological problems. Studies in the literature show that anxiety is positively related to depression, chronic illnesses, career indecision and anxiety. Another variable that anxiety is associated with is perceived stress. Stress is defined as an emotional state that occurs as a result of the perception and evaluation of potential harm in deteriorating living conditions related to the physical and psychological health status of the organism. When environmental demands are perceived to exceed their coping abilities, individuals label themselves as stressed, and in turn, accompanying negative emotional reactions occur. Studies have shown that exposure to chronic stress can lead to the development of various affective disorders, primarily anxiety. When the literature is examined, studies investigating musculoskeletal pain in university students indicate that university students complain most frequently of pain in the spine region, and that low back and neck pain reduce their quality of life in physical, psychological and social aspects. University students are vulnerable to sleep disorders due to environmental reasons such as increased academic stress, anxiety about the future, and increased time spent studying or on extracurricular activities. These reasons are associated with a decrease in total sleep time and deterioration in sleep quality. In studies conducted with university students in Turkey, it has been stated that more than half of the students have poor sleep quality, however, sleep quality is positively related to mental health and physical activity levels. Considering the benefits of physical activity, individuals should be encouraged to engage in physical activity at the most appropriate level for healthier individuals and healthier societies, and it is argued that this is necessary for extending life expectancy and quality of life. When it comes to physical activity and healthy living, yoga comes to mind; It has been interpreted as the process of harmonizing the body with the mind and soul, physically and mentally. In addition, it is stated that yoga practice increases body flexibility, reduces body pain by relaxing muscles, regulates breathing, reduces heart rate, blood pressure and cortisol levels, and reduces stress and anxiety. In addition, regular practice of yoga establishes natural harmony and functional balance between organ systems, making the person feel healthier both physically and mentally. COVID-19, which caused serious respiratory damage in China in the last days of December 2019, has negatively affected not only those infected but also people from all walks of life who have been confined to their homes due to quarantine practices, both physically and psychologically. It has caused congestion in healthcare institutions and difficulties in the provision of healthcare services. For this reason, COVID-19 has increased interest in web-based applications such as telehealth/telemedicine or telerehabilitation. This situation has affected yoga practices, as it has many types of physical activity. In studies comparing face-to-face yoga classes with telehealth yoga classes, it has been reported that similar results were obtained in anxiety and depression levels and that participants were equally satisfied with both methods. In the literature review conducted in light of all this information, no study was found that aimed to develop awareness and well-being through tele-yoga practice for university students with low physical activity levels and experiencing musculoskeletal pain. The aim of this study is to investigate the effects of the tele-yoga program on pain, functionality, anxiety, stress and sleep quality in university students with low physical activity levels and experiencing musculoskeletal pain. In addition, encouraging physical activity in university students and raising awareness, and ensuring holistic well-being in physical, mental and spiritual health are among the goals of the study.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18-26 with low physical activity levels
* Volunteers willing to participate in the study

Exclusion Criteria:

* Individuals with uncontrolled chronic diseases
* Individuals diagnosed with congenital or acquired musculoskeletal disorders or deformities
* Individuals who are currently employed
* Individuals with cardiovascular and/or pulmonary diseases

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline and week 4
  It was used to measure perceived stress in students. The scale contains 10 items on a 5-point Likert scale. Four items are reverse coded and the scale gives a total score. Higher scores indicate higher levels of stress.
Beck Anxiety Inventory (BAI) | Baseline and week 4
  The "Beck Anxiety Scale" was used to question the prevalence of depressive symptoms. The scale measures physical, emotional, and cognitive symptoms of depressive states. The scale includes 21 symptoms based on self-assessment. The highest score that can be obtained is 63; 0-9 points are considered minimal depressive symptoms, 10-16 points are considered mild depressive symptoms, 17-29 points are considered moderate depressive symptoms, and 30 points and above are considered severe depressive symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and week 4
  It was used to measure the sleep quality of the participants.
Perceived Well-Being Scale | Baseline and week 4
  Perceived well-being is the idea that people have about their own health. This idea is usually related to how a person finds themselves (healthy or unhealthy) rather than a true description of their health. In this context, it was used to measure participants' perceptions of well-being.
SF 36 Short Form Questionnaire | Baseline and week 4
  "Short Form-36 (SF-36)" will be used to question the quality of life. SF 36 is a self-assessment scale and examines 8 dimensions of health such as physical function, social function, role limitations (due to physical and emotional reasons), mental health, vitality (energy), pain and general perception of health with 36 items.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda YILDIZ, PhD(c), PT, Principal Investigator — Istanbul Health and Technology University
Locations (1):
- Istanbul Health and Technology University, Istanbul, Beyoğlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No